CLINICAL TRIAL: NCT01246674
Title: Thigh Swelling, Hip-muscle Strength, and Functional Performance Following Total Hip Arthroplasty Monitored Pre-operatively, on the Day of Discharge, and One Week Post-surgery
Brief Title: Thigh Swelling, Hip-muscle Strength, and Functional Performance Following Total Hip Arthroplasty
Acronym: THA
Status: Completed | Type: Observational
Sponsor: Hvidovre University Hospital (Other)
Collaborators: Lundbeck Foundation (Other)
Responsible Party: Principal Investigator, Bente Holm, Physiotherapist for development and research, Hvidovre University Hospital
Other Study IDs: H-4-2010-FSP; THA-BH2 (Registry Identifier: H-4-2010-FSP)
Record Dates: First submitted 2010-11-22; First posted 2010-11-23 (Estimated); Last update posted 2012-07-19 (Estimated); Status verified 2012-07

CONDITIONS: Osteoarthrosis Patients With Total Hip Arthroplasty
Keywords: function, hip muscle strength, hip replacement, hip pain,

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Hypothesis generating study: Consecutive total hip arthroplasty patients

SUMMARY:
By this study the investigators wish to (1) quantify hip strength and functional-performance deficits at discharge after fast-track total hip arthroplasty (THA), and (2) investigate if changes in thigh circumferences, or hip pain are correlated to changes in hip strength and functional-performance after fast-track THA.

DETAILED DESCRIPTION:
The investigators intend to use the results to optimize the rehabilitation programs for THA patients shortly after surgery

ELIGIBILITY:
Inclusion Criteria:

* Total hip arthroplasty patients

Exclusion Criteria:

* inability to speak and understand Danish
* inability to perform the functional measurements due to other conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: from a department of orthopedic surgery
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2011-01; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
hip muscles strength | 6 months

SECONDARY OUTCOMES:
Functional performance | 6 months
  tested by: Timed Up & Go test, 10 meter fast speed walking

CONTACTS AND LOCATIONS:
Overall Officials: Bente Holm, MSc, Principal Investigator — The Lundbeckcenter for hip and knee surgery, University Hospital at Hvidovre, Kettegaard Alle 30, DK-2650 Hvidovre Denmark
Locations (1):
- Dep. of Physical Therapy, Copenhagen University Hospital at Hvidovre, Hvidovre, Hvidovre, Denmark

REFERENCES:
- [Background] Holm B, Kristensen MT, Bencke J, Husted H, Kehlet H, Bandholm T. Loss of knee-extension strength is related to knee swelling after total knee arthroplasty. Arch Phys Med Rehabil. 2010 Nov;91(11):1770-6. doi: 10.1016/j.apmr.2010.07.229. PMID 21044725
- [Derived] Holm B, Thorborg K, Husted H, Kehlet H, Bandholm T. Surgery-induced changes and early recovery of hip-muscle strength, leg-press power, and functional performance after fast-track total hip arthroplasty: a prospective cohort study. PLoS One. 2013 Apr 16;8(4):e62109. doi: 10.1371/journal.pone.0062109. Print 2013. PMID 23614020